CLINICAL TRIAL: NCT03071406
Title: A Phase 2, Randomized, Multi-institutional Study of Nivolumab and Ipilimumab Versus Nivolumab, Ipilimumab and Stereotactic Body Radiation Therapy for Metastatic Merkel Cell Carcinoma
Brief Title: Randomized Study of Nivolumab+Ipilimumab+/- SBRT for Metastatic Merkel Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18786; CA209-737 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2017-03-01; First posted 2017-03-06 (Actual); Results first posted 2023-05-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Merkel Cell Carcinoma; Skin Cancer
Keywords: Merkel cell carcinoma (MCC); Metastatic; Metastasis; Stereotactic body radiation therapy (SBRT); Immunology; Antibody; Nivolumab; Ipilimumab; Metastatic skin cancer; Cutaneous
MeSH Terms: conditions — Carcinoma, Merkel Cell; Skin Neoplasms; Neoplasm Metastasis | interventions — Nivolumab; Ipilimumab; Radiosurgery

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned in a 1:1 ratio to Arm A (nivolumab + ipilimumab), or Arm B (nivolumab + ipilimumab + SBRT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Nivolumab + Ipilimumab (Active Comparator): Nivolumab every 2 weeks and Ipilimumab every 6 weeks until progression or unacceptable toxicity.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Arm B: Nivolumab + Ipilimumab + SBRT (Active Comparator): Nivolumab every 2 weeks and Ipilimumab every 6 weeks until progression or unacceptable toxicity. Stereotactic Body Radiation Therapy (SBRT) to be given at the start of week 2.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 240 mg/dose intravenously (IV) every 2 (q2) weeks.
  Other Names: OPDIVO
Drug: Ipilimumab — Ipilimumab 1 mg/kg/dose IV q6 weeks.
  Other Names: YERVOY
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Stereotactic Body Radiation Therapy 24Gy in 3 fractions.
  Other Names: SBRT
  Arms: Arm B: Nivolumab + Ipilimumab + SBRT

SUMMARY:
The purpose of this study is to test the effectiveness, safety, and tolerability of the drugs nivolumab plus ipilimumab with or without the addition of stereotactic body radiation therapy (SBRT). Nivolumab is an antibody (a type of human protein) that is being tested to see if it will stimulate the body's immune system to work against tumor cells. This study will test an investigational use of nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Eastern Cooperative Oncology Group (ECOG) Performance Status less than 2
* Active disease measurable by CT, MRI or clinical exam.
* Prior chemotherapy or immunotherapy will be allowed if new or persistent measurable site(s) of disease are present.
* Prior radiation therapy will be allowed if there is active measurable disease burden.
* Must be either recurrent, unresectable or Stage IV American Joint Committee on Cancer (AJCC) (7th edition) and have histologically confirmed Merkel cell carcinoma with at least 2 distinct lesions in order to be eligible.
* Must have at least 2 distinct lesions as documented by a complete physical examination or imaging studies within 4 weeks prior to randomization. Imaging studies must include a diagnostic CT scan of the involved disease sites and all known sites of resected disease and brain magnetic resonance (MRI) or CT (brain CT allowable if MRI is contraindicated or if there is no known history of resected brain lesions).
* Tumor tissue from the core biopsy or resected site of disease must be provided for biomarker analyses.

Exclusion Criteria:

* History of Grade 3 toxicity or use of infliximab with prior immunotherapy
* Patients with active brain metastasis.
* Active, known, or suspected autoimmune disease. Potential participants with type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll.
* Patients with prior history of non-Merkel cell carcinoma malignancies are excluded except adequately treated basal cell, squamous cell skin cancer, chronic lymphocytic leukemia or other indolent diseases not requiring therapy; adequately treated, with curative intent, cancer from which the patient is currently in complete remission per investigator's judgment; or patients with history of breast cancer and no evidence of disease on hormonal therapy to prevent recurrence and patients with prostate cancer on adjuvant hormonal therapy with undetectable PSA are eligible.
* A condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization. Inhaled or topical steroids are permitted in the absence of active autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2026-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Wuthrick, M.D, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

REFERENCES:
- [Background] Kim S, Wuthrick E, Blakaj D, Eroglu Z, Verschraegen C, Thapa R, Mills M, Dibs K, Liveringhouse C, Russell J, Caudell JJ, Tarhini A, Markowitz J, Kendra K, Wu R, Chen DT, Berglund A, Michael L, Aoki M, Wang MH, Hamaidi I, Cheng P, de la Iglesia J, Slebos RJ, Chung CH, Knepper TC, Moran-Segura CM, Nguyen JV, Perez BA, Rose T, Harrison L, Messina JL, Sondak VK, Tsai KY, Khushalani NI, Brohl AS. Combined nivolumab and ipilimumab with or without stereotactic body radiation therapy for advanced Merkel cell carcinoma: a randomised, open label, phase 2 trial. Lancet. 2022 Sep 24;400(10357):1008-1019. doi: 10.1016/S0140-6736(22)01659-2. Epub 2022 Sep 12. PMID 36108657
- [Derived] Hoogland AI, Brohl AS, Small BJ, Michael L, Wuthrick E, Eroglu Z, Blakaj D, Verschraegen C, Khushalani NI, Jim HSL, Kim S. Quality of life and patient-reported toxicities in patients with advanced Merkel cell carcinoma treated with combined nivolumab and ipilimumab with or without stereotactic body radiation therapy. Cancer Med. 2024 Jul;13(14):e7464. doi: 10.1002/cam4.7464. PMID 39021272
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: Nivolumab + Ipilimumab | Arm B: Nivolumab + Ipilimumab + SBRT
Started | 25 | 25
Completed | 25 | 24
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Nivolumab + Ipilimumab | Arm B: Nivolumab + Ipilimumab + SBRT | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 19 | 21 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 20 | 19 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 25 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 25 | 25 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response
Description: Overall response according to Immunotherapy Response Evaluation Criteria in Solid Tumors (iRECIST) including Complete Response (CR) + Partial Response (PR).
Time Frame: Up to 18 months
Population: Evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab + Ipilimumab | Arm B: Nivolumab + Ipilimumab + SBRT
Number analyzed (Participants) | 25 | 23
Participants | 18 | 12

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Median Progression Free Survival with 95% Confidence Interval. Progression is defined as progressive tumor lesions per immune-related Response Evaluation in Solid Tumors (irRECIST) definition, or appearance of one or more new Merkel cell carcinoma lesions, which can be local or distant in location from the irradiated lesions.
Time Frame: up to 28 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Nivolumab + Ipilimumab | Arm B: Nivolumab + Ipilimumab + SBRT
Number analyzed (Participants) | 25 | 25
months | 27.7 [9.2 to NA] — Not reached: the upper limit of the 95% confidence interval could not be calculated due to an insufficient number of participants with events | 7.6 [2.8 to NA] — Not reached: the upper limit of the 95% confidence interval could not be calculated due to an insufficient number of participants with events

3. Secondary Outcome: Overall Survival (OS)
Description: Median Overall Survival with 95% Confidence Interval. The length of time from the start of treatment until death from any cause.
Time Frame: Up to 30 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Nivolumab + Ipilimumab | Arm B: Nivolumab + Ipilimumab + SBRT
Number analyzed (Participants) | 25 | 25
months | 29.9 [27.7 to NA] — Not reached: the upper limit of the 95% confidence interval could not be calculated due to an insufficient number of participants with events | 16 [11.3 to NA] — Not reached: the upper limit of the 95% confidence interval could not be calculated due to an insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: Adverse events collected from on study date to 100 days after end of treatment (an average of 10.5 months). Survival will be assessed up to 5 years.
Arm/Group | Arm A: Nivolumab + Ipilimumab | Arm B: Nivolumab + Ipilimumab + SBRT
All-Cause Mortality (participants affected / at risk) | 11/25 | 15/25
Serious Adverse Events (participants affected / at risk) | 13/25 | 13/25
Other Adverse Events (participants affected / at risk) | 25/25 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Nivolumab + Ipilimumab (N=25) | Arm B: Nivolumab + Ipilimumab + SBRT (N=25)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Myocarditis-autoimmune (Cardiac disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (3)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
Enterocolitis infection (Infections and infestations) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 3 (5)
Atrial fibrilation (Cardiac disorders) | 2 (2) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Skin Infection (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Gallbladder obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Vocal fold paralysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) — vocal fold paralysis exacerbated by clinical progression of tumor
MRSA (Infections and infestations) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) — secretions due to recent tracheostomy
Insomnia (Psychiatric disorders) | 0 (0) | 1 (2)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Death NOS (General disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Generalized weakness (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Nivolumab + Ipilimumab (N=25) | Arm B: Nivolumab + Ipilimumab + SBRT (N=25)
Fatigue (General disorders) | 19 (37) | 15 (23)
Edema limbs (General disorders) | 7 (9) | 9 (11)
Pain (General disorders) | 6 (6) | 5 (8)
General disorders and administration site conditions - Other (General disorders) | 4 (4) | 2 (4)
Fever (General disorders) | 4 (4) | 1 (2)
Flu like symptoms (General disorders) | 3 (4) | 2 (3)
Infusion related reaction (General disorders) | 2 (3) | 1 (1)
Chills (General disorders) | 2 (2) | 0 (0)
Localized edema (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Death NOS (General disorders) | 0 (0) | 1 (1)
Edema face (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Irritability (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 10 (21) | 13 (28)
Nausea (Gastrointestinal disorders) | 11 (17) | 10 (12)
Constipation (Gastrointestinal disorders) | 8 (15) | 5 (7)
Abdominal pain (Gastrointestinal disorders) | 4 (7) | 8 (12)
Vomiting (Gastrointestinal disorders) | 4 (4) | 7 (9)
Colitis (Gastrointestinal disorders) | 2 (2) | 8 (12)
Dry mouth (Gastrointestinal disorders) | 3 (4) | 3 (4)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 (2) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Skin lesions (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Actinic Keratoses (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Itching rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Minor rash (Skin and subcutaneous tissue disorders) | 8 (10) | 0 (0)
Macular rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin and subcutaneous tissues disorders - Other (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) — left forearm lesion
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Slight drainage from a couple of the larger lesions with occasional blood tinged discharge from leg lesions
Pruritus (Skin and subcutaneous tissue disorders) | 11 (18) | 10 (15)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (8) | 6 (14)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Weight loss (Investigations) | 8 (12) | 6 (8)
Lipase increased (Investigations) | 7 (15) | 4 (14)
Serum amylase increased (Investigations) | 7 (19) | 4 (8)
Aspartate aminotransferase increased (Investigations) | 7 (21) | 3 (3)
Alanine aminotransferase increased (Investigations) | 6 (35) | 3 (4)
Alkaline phosphatase increased (Investigations) | 3 (3) | 2 (2)
Platelet count decreased (Investigations) | 2 (2) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (2) | 1 (1)
Creatinine increased (Investigations) | 1 (8) | 1 (5)
Weight gain (Investigations) | 1 (2) | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 1 (1)
CPK increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (13) | 11 (14)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 8 (11)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (4)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 12 (14)
Hyponatremia (Metabolism and nutrition disorders) | 7 (12) | 5 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (9) | 4 (5)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 6 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (14) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 2 (4) | 4 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (5) | 0 (0)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (14) | 7 (16)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 6 (12) | 7 (8)
Dizziness (Nervous system disorders) | 5 (6) | 6 (6)
Dysgeusia (Nervous system disorders) | 4 (4) | 2 (2)
Nervous system disorders - Other (Nervous system disorders) | 1 (1) | 2 (3)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1)
Parasthesia (Nervous system disorders) | 1 (2) | 1 (2)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Concentration impairment (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Sinus pain (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (11) | 7 (8) — skin lesion, scheduled for biopsy
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Hypothyroidism (Endocrine disorders) | 5 (5) | 4 (4)
Adrenal insufficiency (Endocrine disorders) | 5 (6) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Endocrine disorders -Other (Endocrine disorders) | 1 (1) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 1 (1) | 0 (0) — Patient reported he has a cold, for which hisPCP treated him with prednisone and amoxicillin
Infections and infestations - Other (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 3 (3)
Wound infection (Infections and infestations) | 1 (1) | 3 (4)
Lung infection (Infections and infestations) | 1 (1) | 2 (2)
Rash pustular (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 6 (11) | 7 (13)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 3 (3) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (3) | 4 (4)
Confusion (Psychiatric disorders) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 4 (6)
Hypertension (Vascular disorders) | 2 (2) | 2 (3)
Lymphedema (Vascular disorders) | 1 (1) | 2 (2)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 2 (3) | 3 (5)
Dry eye (Eye disorders) | 2 (2) | 1 (1)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Stye (Eye disorders) | 0 (0) | 1 (1)
Eye disorders - Other (Eye disorders) | 1 (1) | 0 (0) — Patient reports change in eyesight
Conjunctivitis (Eye disorders) | 1 (1) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 2 (2)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (5)
Hematuria (Renal and urinary disorders) | 2 (3) | 2 (2)
Renal calculi (Renal and urinary disorders) | 2 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 1 (2) | 0 (0)
Heart murmur (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac disorders - Other (Cardiac disorders) | 1 (1) | 0 (0) — Dilated ascending thoracic aorta measures 4.5 cm
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sinus brachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (5) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 4 (5) | 0 (0)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Ear and labyrinth disorders -Other (Ear and labyrinth disorders) | 1 (2) | 0 (0) — Had a sensation and "sound" that there was fluid
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Autoimmune disorder (Immune system disorders) | 1 (1) | 0 (0)
Systemic inflammation syndrome (Immune system disorders) | 0 (0) | 1 (1)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/06/NCT03071406/Prot_SAP_000.pdf